CLINICAL TRIAL: NCT00033813
Title: KUL0401: An Open-label Pilot Study of Oxatomide in Steroid-Naive Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUL0401
Record Dates: First submitted 2002-04-10; First posted 2002-04-11 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne; muscular; dystrophy; controlled clinical trial; CINRG
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — oxatomide

INTERVENTIONS:
Drug: Oxatomide (tinset)

SUMMARY:
This study will help to determine the safety and efficacy of the mast cell stabilizer Oxatomide as a treatment for Duchenne muscular dystrophy (DMD). Boys with DMD who are enrolled in this study will should not have taken steroids to treat DMD for at least twelve months, and should not have taken any nutritional supplements for at least three months. Subjects will complete a two screening visits within a one-week period, and if enrolled will then have their strength tested monthly for three months before beginning therapy with Oxatomide. Once Oxatomide therapy is started, participants will have their strength tested monthly for six months. Following the six month treatment period, participants will be given the option to remain on Oxatomide until the study is completed.

ELIGIBILITY:
Subject Inclusion Criteria

1. 5 to 10 years of age
2. ambulatory
3. diagnosis of DMD confirmed by at least one of the following:

   * Positive x-linked family history of DMD in older male relatives (onset by 5 years, wheelchair bound by 12 years), or;
   * Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical picture consistent with typical DMD, or;
   * Gene deletion test positive (missing one or more exons) in the central rod domain (exons 25-60) of dystrophin, where reading frame can be predicted as 'out of frame', and clinical picture consistent with typical DMD.
4. glucocorticosteroid-naive (i.e. has not been treated with prednisone or deflazacort within the past year)
5. Evidence of muscle weakness by MRC score or clinical functional evaluation
6. QMT biceps score variability no greater than 10% between screening visits

Subject Exclusion Criteria

1. Failure to achieve one or more of the inclusion criteria listed above
2. Inability to suitably cooperate with strength assessments
3. Symptomatic DMD carrier
4. Use of oxatomide (or other anti-histamine drugs) within the last 6 months for DMD or any other disease
5. Use of creatine monohydrate or glutamine within the last 6 months
6. Use of carnitine, Coenzyme Q10, other amino acids or any herbal medications within the last 3 months
7. History of symptomatic cardiomyopathy
8. History of impairment of hepatic function
9. History of significant concomitant illness or significant impairment of renal function.

Ages: 5 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15
Dates: Start 2002-01; Primary Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- See also: The Cooperative International Neuromuscular Research Group — http://www.cnmcresearch.org/cinrg/index.asp